CLINICAL TRIAL: NCT02469844
Title: Heart Rate Variability (HRV) Analysis in Patients With Nocturnal Epileptic Seizures
Status: Completed | Type: Observational
Sponsor: Sheffield Teaching Hospitals NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: STH18174
Record Dates: First submitted 2015-06-03; First posted 2015-06-12 (Estimated); Last update posted 2023-11-15 (Actual); Status verified 2023-11

CONDITIONS: Heart Rate; Nocturnal Seizures; Autonomic Nervous System; Epilepsy
MeSH Terms: conditions — Epilepsy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Patients with epilepsy having seizures in sleep

SUMMARY:
Epilepsy is disabling and costly to patients and the health service. Nearly 400,000 people in England suffer from epilepsy. About 40% of these patients are known to have seizures predominantly in sleep. All seizures pose risk to the individual both physical and psychological. Nocturnal seizures pose extra risk as the diagnosis may be missed or delayed. Patients with nocturnal seizures are also thought to be at particular risk of sudden unexpected death in epilepsy (SUDEP), especially if their seizures are unobserved. In patients with poor seizure control, the risk of SUDEP has been found to be as high as 9 per 1,000 patient years. Previous studies show that many seizures are associated with changes in the Autonomic Nervous System (ANS) tone. The ANS tone can be assessed using heart rate variability parameters (HRV). A few studies suggest that ANS tone changes tend to precede the onset of epileptic seizure related surface electroencephalographic (EEG) changes, suggesting that ANS tone changes could be used in seizure alarm or intervention systems. This prospective study intends to focus on seizures from sleep and study HRV parameters in the immediate preictal state of the seizure and compare these with resting HRV parameters in the same patient with the aim of finding HRV metrics which could help to identify the presence of seizures in longterm electrocardiographic (ECG) recordings, or help predict seizure occurrence, or provide information about the current risk of seizures. This study will also investigate whether there are differences in the alterations of HRV parameters between different forms of epilepsy and whether seizure lateralisation has an impact on HRV parameters.

ELIGIBILITY:
Inclusion Criteria:

1. Clinically firm diagnosis of epilepsy.
2. 18 years of age
3. Having the capacity to consent to this project.

Exclusion Criteria:

1. Patients who are on medication for cardiac conditions like beta blockers, anti arrhythmic agents, calcium channel blockers.
2. Patients who have other neurological disorders which may be associated with an autonomic neuropathy
3. Patients who have diabetes, renal failure or another general medical disorder associated with autonomic neuropathy.
4. Patients unable to complete self-report measures unaided.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with epilepsy admitted for three- to five-day diagnostic or pre-surgery video-electro-encephalography and ECG (VT) monitoring in the video telemetry unit at the Royal Hallamshire Hospital in Sheffield will be recruited for the study.
Sampling Method: Non-Probability Sample
Enrollment: 48 (Actual)
Dates: Start 2014-10 (Actual); Primary Completion 2018-12 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Alterations in heart rate variability (HRV) parameters at baseline (interictal sleep), immediately before (pre-ictal) and during nocturnal epileptic seizures in epilepsy patients. | Alterations in HRV during nocturnal seizures occuring during patients stay in VT unit for 3-5 days
  1. Alterations in heart rate variability (HRV) parameters at baseline (interictal sleep), immediately before (pre-ictal) and during nocturnal epileptic seizures. The composite measure consists of the following: Time Domain HRV metrics: SDNN to describe overall variability; RMSSD to describe Parasympathetic component of HRV FrequencyDomain HRV: HF for Parasympathetic, LF for Sympathetic and LF/HF for sympatho vagal balance.
  Non-linear HRV metrics: CVI for Parasympathetic and CSI for Sympathetic component.

SECONDARY OUTCOMES:
Comparing Alterations in the HRV parameters in temporal lobe epileptic seizures from extra temporal lobe epileptic seizures. | Alterations in HRV during nocturnal seizures occuring during patients stay in VT unit for 3-5 days

CONTACTS AND LOCATIONS:
Overall Officials: Athi Ponnusamy, MD, Principal Investigator — Sheffield Teaching Hospitals NHS Foundation Trust
Locations (1):
- Sheffield Teaching Hospitals NHS Foundation Trust, Sheffield, South Yorkshire, United Kingdom

REFERENCES:
- [Background] Ponnusamy A, Marques JL, Reuber M. Heart rate variability measures as biomarkers in patients with psychogenic nonepileptic seizures: potential and limitations. Epilepsy Behav. 2011 Dec;22(4):685-91. doi: 10.1016/j.yebeh.2011.08.020. Epub 2011 Oct 4. PMID 21975299
- [Background] Ponnusamy A, Marques JL, Reuber M. Comparison of heart rate variability parameters during complex partial seizures and psychogenic nonepileptic seizures. Epilepsia. 2012 Aug;53(8):1314-21. doi: 10.1111/j.1528-1167.2012.03518.x. Epub 2012 May 29. PMID 22642646